CLINICAL TRIAL: NCT04580745
Title: A Phase 1a Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Oral MORF-057 in Healthy Subjects
Brief Title: Study of MORF 057 to Evaluate Single and Multi Ascending Doses in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morphic Therapeutic, Inc. (A Wholly Owned Subsidiary of Eli Lilly and Company) (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 27496; J6E-MC-KWAE (Other: Eli Lilly and Company); MORF-057-101 (Other: Morphic ID)
Record Dates: First submitted 2020-09-16; First posted 2020-10-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: MORF-057

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MORF-057 (Experimental): SAD: Subjects will be assigned to one of five planned dose cohorts and receive single doses of MORF-057.
  Food Effect: Subjects will receive single dose administration of MORF-057 in fed and fasted states.
  MAD: Subjects will be assigned to one of three planned dose cohorts and receive multiple doses of MORF-057.
  Interventions: Drug: MORF-057
- Placebo for MORF-057 (Experimental): SAD: Subjects will be assigned to one of five planned dose cohorts and receive single doses of placebo.
  MAD: Subjects will be assigned to one of three planned dose cohorts and receive multiple doses of placebo.
  Interventions: Drug: Placebo for MORF-057

INTERVENTIONS:
Drug: MORF-057 — SAD: Subjects will be assigned to one of five planned dose cohorts and receive single doses of MORF-057.
  Food Effect: Subjects will receive single dose administration of MORF-057 in fed and fasted states.
  MAD: Subjects will be assigned to one of three planned dose cohorts and receive multiple doses of MORF-057.
  Arms: MORF-057
Drug: Placebo for MORF-057 — SAD: Subjects will be assigned to one of five planned dose cohorts and receive single doses of placebo.
  MAD: Subjects will be assigned to one of three planned dose cohorts and receive multiple doses of placebo.
  Arms: Placebo for MORF-057

SUMMARY:
Phase 1a randomized, double-blind, placebo-controlled study to evaluate single and multiple ascending doses of MORF-057 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 to 65 years old with a body mass index between 18 and 32 kg/m2
* Determined to be medically healthy by the Investigator.
* Use of acceptable methods of contraceptives.
* Ability to provide written informed consent and to understand and comply with the requirements of the study.

Exclusion Criteria:

* History of any malignancy, except basal or squamous cell carcinoma of the skin that resolved or in remission prior to Screening.
* Abnormal laboratory values at Screening.
* Any clinically significant major diseases.
* Female who is pregnant or breastfeeding, or planning to become pregnant during the course of the study.
* Unwilling or unable to comply with the requirements of the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and safety signals observed during single and multiple ascending doses of MORF-057 administered orally to healthy adult subjects | Day -1 to Day 28
  Subject incidence of adverse events and serious adverse events
Maximum Plasma Concentration (Cmax) of MORF-057 in a fed state | Day -1 to Day 28
  Cmax (Food Effect cohort)
Time to Reach Cmax (Tmax) of MORF-057 in a fed state | Day -1 to Day 28
  Tmax (Food Effect cohort)

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) during single and multiple ascending doses of MORF-057 | Day -1 to Day 28
  Cmax of MORF-057
Time to Reach Cmax (Tmax) during single and multiple ascending doses of MORF-057 | Day -1 to Day 28
  Tmax of MORF-057
Incidence of adverse events and safety signals observed during single dose of MORF-057 administered after a meal to healthy subjects. | Day -1 to Day 28
  Subject incidence of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace, Cincinnati, Ohio, United States